CLINICAL TRIAL: NCT02511951
Title: A Prospective Randomized Clinical Trial of Two Surgical Techniques for Pancreaticojejunostomy in Patients Undergoing Pancreaticoduodenectomy: One-layer Versus Two-layer Duct-to-mucosa Pancreaticojejunostomy
Brief Title: One-layer Versus Two-layer Duct-to-mucosa Pancreaticojejunostomy After Pancreaticoduodenectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Anhui Medical University (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, xpgeng, vice-president, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ahykdxdefsyy11
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Pancreatic Fistula
Keywords: postoperative pancreatic fistula; postoperative hospital stay time; anastomosis time; reoperation rate; morbidity; pancreaticojejunostomy; pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Fistula | interventions — Pancreaticojejunostomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- one-layer duct-to-mucosa anastomosis (Experimental): one-layer duct-to-mucosa anastomosis is used for pancreaticojejunostomy after pancreaticoduodenectomy.
  Interventions: Procedure: pancreaticojejunostomy
- two-layer duct-to-mucosa anastomosis (Active Comparator): two-layer duct-to-mucosa anastomosis is used for pancreaticojejunostomy after pancreaticoduodenectomy.
  Interventions: Procedure: pancreaticojejunostomy

INTERVENTIONS:
Procedure: pancreaticojejunostomy — To create the posterior suturing layers, the needle is inserted from the posterior interior side of the pancreatic duct, passing through the dorsal region of the parenchyma of the pancreatic stump to the posterior surface of the pancreas approximately 0.5 cm distal to the cut edge. The other side of the needle starts from the inside of the jejunum lumen to the subserosa and then passes through the seromuscular layer to the posterior surface of the bowel.The anterior suturing layer is performed in the same manner.
  Two layer anatomosis with "Duct-to-Mucosa" pancreaticojejunostomy is performed by suturing the pancreatic parenchyma to the jejunal seromuscular layer and no stenting tube was used.

SUMMARY:
The aim of this study is to investigate a new pancreaticojejunal (PJ) anastomosis procedure named "One-layer duct-to-mucosa pancreaticojejunostomy" in pancreatoduodenectomy, which could provide a feasible option to pancreatic surgeons for patients with pancreaticoduodenectomy.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy is a standard surgical approach for resectable pancreatic tumors and periampullary tumors. It is considered a safe procedure resulting from the continuous improvement in surgical techniques over the years. Although postoperative mortality has obviously decreased, pancreatic fistula is still a major challenge in pancreatic surgery and remains the major cause of postoperative morbidity and mortality after pancreaticoduodenectomy(PD), ranging from 3% to 30%.

Many risks factors have been shown to cause pancreatic fistula(PF) after the operation, including advanced age, prolonged operation time, intraoperative hemorrhage, BMI, soft pancreas, size of the main pancreatic duct and texture of the remnant pancreas. Among them, soft pancreatic texture without a dilated main pancreatic duct is regarded as the most important risk factor in predicting pancreatic fistula.

The serious consequences of pancreatic fistula result from the pancreatic juice becoming activated by the bile and intestinal fluid, which will eventually corrupt the PJ anastomosis and the surrounding normal tissues. The corrosion of the vasculature will lead to lethal hemorrhage, which is the main cause of mortality after pancreaticoduodenectomy. Furthermore, pancreatin, together with the bacteria in the alimentary tract, will lead to intra-abdominal infection and abscess. To reduce the pancreatic fistula rate, several techniques have been described as alternatives to the conventional PJ anastomosis. Duct-to-mucosa sutures, binding pancreaticojejunostomy and end-to-side invaginated fashion are widely used in the current clinical setting. Some non-randomized studies showed that the one-layer duct-to-mucosa method was a relatively safe approach. However, the prospective clinical study found that in comparison with the conventional two-layer duct-to-mucosa did obviously decrease the incidence of pancreatic fistula as well as other operative complications. The postoperative pancreatic fistula (POPF), which determines postoperative mortality, length of hospital stay， is dependent of its definition, and is reported in up to 16% of patients. The purpose of this study is to determine whether the new anastomosis called " one-layer duct-to-mucosa " pancreaticojejunostomy can reduce the POPF rate and downgrade compared with the common accepted duct-to-mucosa pancreaticojejunostomy after pancreaticoduodenectomy. This single-centre, open, randomized controlled trail is conducted following International Study Group on Pancreatic Fistula (ISGPF) criteria for pancreatic fistula (PF). The primary endpoint is the POPF rate, and others include overall postoperative complication rate and their severity reoperation rate and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female, aged 18 to 80;
* Patients scheduled to undergo pancreaticoduodenectomy;
* Provided written informed consent;

Exclusion criteria:

* Patients with severe cardiopulmonary disorder that might prolong the postoperative hospital stay;
* Patients who had a previous pancreatic operation;
* Patients with an immunodeficiency;
* Patients who underwent an emergency operation;
* Pregnant patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
postoperative pancreatic fistula(POPF) rate | 30 days
  drainage of any measurable volume of fluid with an amylase content >3 times the upper normal serum value on or after postoperative day 3.

SECONDARY OUTCOMES:
Duration of postoperative hospital stay | 30 days
  Time from day of operation to day of discharge
anastomosis time | 1 hour
  anastomosis time was calculated from begining to the end of pancreaticojejunostomy
reoperation rate | 30 days
  The secondary endpoint will be the reoperation rate
Morbidity | 30 days
  the severity of complications was graded according to the Clavien-Dindo classification
Mortality | 30 days
  operative mortality was defined as any death resulting from a complication during surgery
Biliary leakage | 30
  biliary leakage was documented in line with the International Study Group of Liver Surgery(ISGLS) definitions and grading systems
Blood transfusion | 2 days
  Administration of blood transfusions is documented for the intraoperative and postoperative period until 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: xiaoping geng, professor, Principal Investigator — the vice President of the second affiliated hospitalof Anhui medical university
Locations (1):
- the Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Result] Zhang L, Li Z, Wu X, Li Y, Zeng Z. Sealing pancreaticojejunostomy in combination with duct parenchyma to mucosa seromuscular one-layer anastomosis: a novel technique to prevent pancreatic fistula after pancreaticoduodenectomy. J Am Coll Surg. 2015 May;220(5):e71-7. doi: 10.1016/j.jamcollsurg.2014.12.047. Epub 2015 Jan 15. No abstract available. PMID 25840535
- [Result] Wei J, Liu X, Wu J, Xu W, Zhou J, Lu Z, Chen J, Guo F, Gao W, Li Q, Jiang K, Dai C, Miao Y. Modified One-layer Duct-to-mucosa Pancreaticojejunostomy Reduces Pancreatic Fistula After Pancreaticoduodenectomy. Int Surg. 2015 Jun 3. doi: 10.9738/INTSURG-D-15-00094.1. Online ahead of print. PMID 26037262
- [Result] El Nakeeb A, El Hemaly M, Askr W, Abd Ellatif M, Hamed H, Elghawalby A, Attia M, Abdallah T, Abd ElWahab M. Comparative study between duct to mucosa and invagination pancreaticojejunostomy after pancreaticoduodenectomy: a prospective randomized study. Int J Surg. 2015 Apr;16(Pt A):1-6. doi: 10.1016/j.ijsu.2015.02.002. Epub 2015 Feb 13. PMID 25682724
- [Derived] Pan SB, Geng W, Zhou DC, Chen JM, Zhao HC, Liu FB, Xie SX, Hou H, Zhao YJ, Xie K, Wang GB, Geng XP. One-layer versus two-layer duct-to-mucosa pancreaticojejunostomy after pancreaticoduodenectomy: study protocol for a randomized controlled trial. Trials. 2016 Aug 17;17(1):407. doi: 10.1186/s13063-016-1517-8. PMID 27530630